CLINICAL TRIAL: NCT00697554
Title: Study to Compare the Immunogenicity and Safety of GSK Biologicals' Novel Adjuvanted HBV Vaccine (0, 21-day Schedule) to a Double Dose of Engerix™ -B (0, 7, 21-day Schedule), in Pre-liver Transplant Patients ≥ 18 y, Boosted at Month 6-12
Brief Title: Immunogenicity and Safety of a Novel Adjuvanted HBV Vaccine in Pre-liver Transplant Patients 18 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/036
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Adjuvanted hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: HBV-MPL vaccine 208129
- Group B (Active Comparator)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBV-MPL vaccine 208129 — 2-dose primary vaccination followed by 1 booster vaccination by intramuscular injection
  Arms: Group A
Biological: Engerix™-B — 3-dose primary vaccination followed by 1 booster vaccination by intramuscular injection of double doses
  Other Names: HBV-MPL vaccine 208129
  Arms: Group B

SUMMARY:
The purpose of this study is to enroll pre-liver transplant patients who will be vaccinated with either the novel adjuvanted HBV vaccine or double doses of Engerix™-B. The immunogenicity and safety of the novel adjuvanted vaccine will be compared to Engerix™-B as the control vaccine

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* A male or female ≥ 18 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Seronegative for anti-HBs-antibodies, anti-HBc-antibodies & HBsAg.
* If the subject is female, she must be of non-childbearing potential or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.
* Documented case of liver failure, such that the patient will require an eventual liver transplant

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days preceding the first dose of study vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of vaccine and ending 30 days after.
* Previous vaccination against hepatitis B (whether or not a non-responder to vaccination).
* Previous vaccination with an adjuvant system containing MPL®.
* History of hepatitis B infection.
* Known exposure to hepatitis B virus within 6 weeks.
* Previously confirmed human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* Immunosuppression caused by the administration of parenteral steroids or chemotherapy.
* Suspected or confirmed multiple sclerosis in the subject (applicable to Centres 011, 012, 013 and 014/ France only).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute, intercurrent disease at the time of enrollment.
* Oral/axillary temperature of ≥ 37.5°C (≥ 99.5°F).
* Administration of immunoglobulins and/or any blood products within one month preceding the first dose of study vaccine or planned administration/ administration during the study period.
* Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2000-01; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | At Day 28

SECONDARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of solicited local and general signs and symptoms | During a 4 day follow-up period after vaccination
Occurrence, intensity and relationship to vaccination of unsolicited symptoms | During a 30 day follow-up period after vaccination
Occurrence, intensity and relationship to vaccination of serious adverse events (SAEs) | During the study period
Anti-HBs antibody concentrations | At d21, d28, d56, M6-12, 1M after booster dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nevens F, Zuckerman JN, Burroughs AK, Jung MC, Bayas JM, Kallinowski B, Rivas EF, Duvoux C, Neuhaus P, Saliba F, Buti M, Zarski JP, Pons F, Vanlemmens C, Hamtiaux V, Stoffel M. Immunogenicity and safety of an experimental adjuvanted hepatitis B candidate vaccine in liver transplant patients. Liver Transpl. 2006 Oct;12(10):1489-95. doi: 10.1002/lt.20836. PMID 16964595
- [Background] Nevens F et al. Immunogenicity and safety of a novel adjuvanted hepatitis B candidate vaccine in liver transplant patients. Abstract presented at the 39th Annual Meeting of the European Association for the Study of Liver (EASL), Berlin, Germany, 14-18 April 2004.
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 208129/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208129/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208129/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208129/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208129/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register